CLINICAL TRIAL: NCT05845944
Title: Evaluation of the Efficiency of the Video-supported Education Given to Students for Nasogastric Tube Feeding in Pediatric Patient
Brief Title: Video Education About Nasogastric Tube Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, Şeyda BİNAY YAZ, Assistant professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Bakircay1
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Nutrition, Healthy; Nurse's Role; Education; Pediatric
Keywords: Nursing students; Education; Pediatric patient; Nasogastric tube; Feeding

STUDY DESIGN:
Intervention Model Description: The research was a randomized controlled, experimental study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-supported education group (Experimental): All participants in this group were given the "Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients" prepared by the researchers as a pre-test.
  The participants of this group, who were determined by randomization, were given education prepared using the video-supported education method. The education took 35 minutes. After the training, the "Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients" was applied as a post-test.
  Interventions: Other: Video-supported education group
- Control Group (No Intervention): No intervention was made. All participants in this group were given the "Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients" prepared by the researchers as a pre-test.
  Afterward, theoretical information on the subject was given. After theoretical information, the "Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients" was applied as a post-test.

INTERVENTIONS:
Other: Video-supported education group — Providing training on nutrition with a nasogastric tube in pediatric patients with a video-supported education method
  Arms: Video-supported education group

SUMMARY:
Summary Aim: This research was conducted to determine the effectiveness of education given to students using video in feeding with the nasogastric tube for pediatric patients.

Method: It was a randomized controlled experimental study. The sample of the study consisted of 61 nursing students. The students included in the study were divided into two equal groups: the experimental and control groups. Video-supported education material of the experimental group and theoretical education was applied to the control group. Before and after the education, a post-knowledge test was made and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of the Department of Nursing
* Taking the child health and diseases nursing course and being successful
* Volunteering to participate in the research

Exclusion Criteria:

* Participate and quit the study
* Being a 1st and 2nd year nursing student
* Failure of the child health and diseases nursing course

Ages: 19 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Statistical difference between groups about knowledge test scores | During the education, approximately 35 minutes
  Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients was applied twice as a pre-test and post-test in experimental and control groups. Knowledge Test on Nasogastric Tube Feeding in Pediatric Patients: It is a 17-question form prepared by researchers. Content validity has been made for the form. Each correct answer is calculated as 1 point and each wrong answer is calculated as 0 points. The higher the score obtained from the questionnaire, the higher the level of knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Atay, Principal Investigator — Izmir Bakircay University
Locations (1):
- Bakırcay University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study will be prepared for publication